CLINICAL TRIAL: NCT05268666
Title: A First-in-Human, Open-label, Dose Escalation and Expansion Study of Orally Administered JBI-802 in Patients With Advanced Solid Tumors
Brief Title: A Study of Orally Administered JBI-802, an LSD1/HDAC6 Inhibitor, in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jubilant Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JBI-802-101
Record Dates: First submitted 2022-02-11; First posted 2022-03-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-08

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: SCLC; neuroendocrine prostate cancer; neuroendocrine; JBI-802
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JBI-802 (Experimental): 10 mg JBI-802 once daily as the starting dose with 4 days on/3 days off cycle
  Interventions: Drug: JBI-802

INTERVENTIONS:
Drug: JBI-802 — LSD1/HDAC6 inhibitor

SUMMARY:
The purpose of this study is to determine the maximum-tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of JBI-802 in patients with Advanced Solid Tumors.The efficacy of the RP2D will be evaluated in phase 2 in patients with solid tumors of neuroendocrine differentiation.

DETAILED DESCRIPTION:
This is a multi-center, first in human, open-label, 2-part, dose escalation and expansion study to define safety, tolerability, maximum tolerated dose, pharmacologically active dose, assess preliminary efficacy, and explore predictive and pharmacodynamic biomarkers in up to 126 participants with advanced solid tumors. Expansion cohorts of participants, treated at the RP2D, with small cell lung cancer (SCLC), neuroendocrine prostate cancer (NEPC), and other neuroendocrine-derived cancers will be enrolled to obtain additional safety and efficacy data. Starting dose will be 10 mg orally once daily, 4 days on and 3 days off cycle.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years at Screening
* Absolute neutrophil count (ANC) ≥1500 cells/mm3.
* Platelet count ≥100,000 cells/mm3.
* Total bilirubin ≤1.5×ULN. Patients with Gilbert's syndrome may be enrolled with up to 3.0xULN.
* AST and ALT ≤2.5×ULN (unless liver metastases are present then up to 5×ULN is allowed).
* Calculated creatinine clearance (CrCL) ≥60 mL/min (Cockcroft-Gault formula).
* Prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN if participant is not anticoagulated (Note: If participant is on anticoagulants, the participant must be on a stable dose for at least 2 weeks prior to study entry.
* Must have at least one measurable lesion on CT scan or MRI per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Other criteria may apply

Part 1:

* Participants with a histologically confirmed diagnosis of locally advanced or metastatic solid tumors (except microsatellite stable colorectal cancer and hepatocellular carcinoma) who have no available effective therapeutic options.

Part 2:

* Small cell lung cancer: Participants must have a histologic diagnosis of advanced SCLC not amenable to curative therapy and have received ≤2 prior regimens, which must have included a checkpoint inhibitor and a platinum-based chemotherapy.
* De novo or treatment-emergent NEPC
* Basket of neuroendocrine-derived tumors, excluding SCLC and treatment-induced NEPC. Participants must have unresectable locally advanced or metastatic disease and have no available effective therapeutic options.

Exclusion Criteria:

* Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or hemorrhage for at least 4 weeks after treatment (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of symptomatic brain metastases for at least 14 days prior to enrollment.
* Severe or unstable medical condition, such as congestive heart failure (New York Heart Association [NYHA] Class III or Class IV), ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, as well as an uncontrolled cardiac arrhythmia requiring medication (≥Grade 2, according to NCI CTCAE Version 5), myocardial infarction within 6 months prior to starting study treatment, or any other significant or unstable concurrent cardiac illness. Note: Stable chronic atrial fibrillation is allowed.
* Use of strong inhibitors of CYP3A within 14 days or 5 half-lives (whichever is longer) or grapefruit juice or grapefruit containing products within 7 days prior to Cycle 1 Day 1.
* Use of strong inducers of CYP3A within 14 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
* Use of strong inhibitors of cytochrome CYP2D6 within 14 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
* Use of strong inducers of CYP2D6 within 14 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
* History of other previous or concurrent cancer that would interfere with the determination of safety or efficacy assessment
* Surgery (eg, stomach bypass) or medical condition that might significantly affect absorption of medicines
* Other criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Maximum-Tolerated Dose (MTD) | 28-day cycle
Investigator-Assessed ORR (Part 2) | Up to 30 days from the last dose of study drug
  Defined as either complete response (CR) or partial response (PR) as defined by RECIST version 1.1

SECONDARY OUTCOMES:
Incidence of AEs | Up to 30 days from the last dose of study drug
  Characterized overall and by type, seriousness, relationship to study treatment, timing, and severity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Cmax: Maximum Plasma Concentration JBI-802 | Baseline up to 28 days from the last dose of study drug
  Defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations.
Tmax: Time of Maximum Plasma Concentration JBI-802 | Baseline up to 28 days from the last dose of study drug
  Defined as the time at which the Cmax occurs.
Clast: Last Observed (quantifiable) Plasma Concentration in units of ng/mL JBI-802 | Baseline up to 28 days from the last dose of study drug
  Last Observed (quantifiable) Plasma Concentration in units of ng/mL JBI-802
AUC(0-last): Area Under the Concentration-time Curve from Dosing (time 0) to Time of Last Measured Concentration JBI-802 | Baseline up to 28 days from the last dose of study drug
  AUCs will be reported in units of h×ng/mL
AUC(0-t) (partial AUC): Area Under the Concentration-time Curve from Dosing (time 0) to Time t JBI-802 | Baseline up to 28 days from the last dose of study drug
  May be computed for one or more values of t, with specific values of t determined after observing the data; AUCs will be reported in units of h×ng/mL
Vd/F: Apparent Volume of Distribution During Terminal Phase (Vz/F) After Oral Administration calculated as (CL/F)/ Ke | Baseline up to 28 days from the last dose of study drug
  Volume will be reported in units of L.
CL/F: Apparent Oral Clearance (CL/F) computed as Dose/AUC | Baseline up to 28 days from the last dose of study drug
  Clearance will be reported in units of L/h.
t½: The Apparent Terminal Elimination Half-life JBI-802 | Baseline up to 28 days from the last dose of study drug
  The time required for the drug concentration to decrease by a factor of one-half in the terminal phase. t½ can be estimated as ln(2) / Ke. t1/2 will be reported in units of h.
Investigator-Assessed Overall Response Rate (ORR) (Part 1) | Up to 30 days from the last dose of study drug
  ORR is defined as the percentage of patients with a confirmed complete response (CR) or a partial response based on RECIST 1.1
Duration of Response (DOR) | Up to 30 days from the last dose of study drug
  Time from the date of first documented CR or PR, assessed by the investigator and based on RECIST 1.1 to the documented date of progressive disease (PD) or death, whichever occurred first
PFS: Progression Free Survival | Date patient started study drug to date of progression, assessed up to 30 months
  The time from the date the patient started study drug to the date the patient experiences an event of disease progression
OS: Overall Survival | Date patient started study drug to date of death for any cause, assessed up to 30 months
  The time from the date patient started study drug to death for any reason
PSA 50 Response Rate in Patients with Prostate Cancer | Baseline up to 30 days from the last dose of study drug
  The percentage of patients who experience a ≥50% decline in PSA from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Program Manager, Study Director — Jubilant Therapeutics Inc.
Locations (4):
- United States (4):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - The Christ Hospital, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - NEXT Virginia, LLC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No